CLINICAL TRIAL: NCT05049343
Title: A Phase 1, Double-Blind, Placebo-Controlled Crossover Study of SAGE-904 Using a Ketamine Challenge to Evaluate Electrophysiology, Safety, Tolerability, and Pharmacokinetics in Healthy Participants
Brief Title: Study of SAGE-904 Using a Ketamine Challenge to Evaluate Electrophysiology, Safety, Tolerability, and Pharmacokinetics in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 904-TRM-101
Record Dates: First submitted 2021-09-10; First posted 2021-09-20 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; SAGE-904; Ketamine
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SAGE-904 then Placebo (Experimental): SAGE-904 in combination with ketamine, followed by a washout period, followed by placebo in combination with ketamine.
  Interventions: Drug: SAGE-904; Drug: Placebo; Drug: Ketamine
- Placebo then SAGE-904 (Placebo Comparator): Placebo in combination with ketamine, followed by a washout period, followed by SAGE-904 in combination with ketamine.
  Interventions: Drug: SAGE-904; Drug: Placebo; Drug: Ketamine

INTERVENTIONS:
Drug: SAGE-904 — SAGE-904 oral solution.
Drug: Placebo — Placebo oral solution.
Drug: Ketamine — Ketamine intravenous (IV) infusion.

SUMMARY:
The primary purpose of this study is to determine functional target engagement of SAGE-904 using electrophysiological paradigms before and after ketamine administration.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to provide 2 forms of identification; at least 1 must have a photo
2. Participant has a body weight ≥50 kilograms (kg) and body mass index ≥18.0 and ≤30.0 kilograms per square meter (kg/m^2) at screening
3. Participant is healthy with no history or evidence of clinically relevant medical disorders as determined by the investigator
4. Participant has the ability to tolerate the electrode headset for the duration of the testing session

Exclusion Criteria:

1. Participant has a history or presence of any psychiatric disease or condition including suicidal ideation or behavior, has answered YES to any question on the Columbia-Suicide Severity Rating Scale (C-SSRS) at screening or admission, or is currently at risk of suicide in the opinion of the Investigator
2. Participant has a history or presence of a neurologic disease or condition, including, but not limited to, epilepsy, closed head trauma with clinically significant (CS) sequelae, or a prior seizure
3. Participant has a family history of epilepsy
4. Participant has a history, presence, and/or current evidence of serologic positive results for Hepatitis B and C, human immunodeficiency virus (HIV) 1 or 2
5. Participant has obstructed venous access and/or has skin disease, rash, acne, or abrasion at venous access site that may affect the ability to obtain a pharmacokinetic (PK) sample or affect the ability to receive the ketamine infusions
6. Participant has had previous exposure to or is known to be allergic to ketamine or any of its excipients

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Change in Electrophysiological Parameter: Auditory Evoked Potential (AEP) in a Single-stimulus Paradigm Before and After Ketamine Infusion in Participants Receiving SAGE-904 Versus (vs) Participants Receiving Placebo | Pre-dose and post-dose on Days 1 and 11
  AEP variables will include individual amplitudes of N100 and P200 responses and the derived peak-to-peak amplitude of these responses (N100-P200) in microvolts (µV).
Change in Electrophysiological Parameter: Mismatch Negativity (MMN) Before and After Ketamine Infusion in Participants Receiving SAGE-904 vs Participants Receiving Placebo | Pre-dose and post-dose on Days 1 and 11
  MMN is a response to nonmatching sounds in a series of matching sounds. Two tones of the same frequency and sound intensity, but differing in duration, will be sequentially presented to the participant through insert earphones. MMN amplitude will be measured from the peak of a mid-latency negative voltage deflection in the difference waveform representing the response to deviant stimuli in µV.
Change in Electrophysiological Parameter: Auditory Steady-state Response (ASSR) Power Before and After Ketamine Infusion in Participants Receiving SAGE-904 vs Participants Receiving Placebo | Pre-dose and post-dose on Days 1 and 11
  ASSR is used to assess the integrity of sensory pathways including cortical processing. ASSR will be measured at midline central electrode (Cz) of electroencephalogram (EEG) to assess the response in hertz (Hz). In ASSR, streams of "click" stimuli will be presented at a rate of 40 Hz while the participant will be instructed to fix their gaze on a white cross displayed on a computer monitor.
Change in Electrophysiological Parameter: P300 in a Target Detection Paradigm as Assessed by Auditory Response Before and After Ketamine Infusion in Participants Receiving SAGE-904 vs Participants Receiving Placebo | Pre-dose and post-dose on Days 1 and 11
  Improvement of the P300 auditory response time in milliseconds using P300 AEP in a target detection paradigm by an increase in amplitude and/or a decrease in latency will be analyzed. In this paradigm, 2 tones of the same sound intensity, but differing in frequency, are sequentially presented to the participant through insert earphones. The "standard" (low frequency) stimuli will be presented on the majority of trials, with a "target" (high frequency) stimuli presented periodically at random. The participant is told to listen for the "target" stimuli and press a button on the handset as fast as they can. The endpoint variables of P300 amplitude and latency in correlation with the button press reaction time will be used to assess the response time.

SECONDARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Up to Day 25
  An adverse event (AE) is any untoward medical occurrence in a patients or clinical investigation participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. A TEAE is defined as an AE with onset after the start of investigational product (IP), or any worsening of a pre-existing medical condition/AE with onset after the start of IP and throughout the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Sage Investigational Site, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.